CLINICAL TRIAL: NCT01584908
Title: Adjuvanted Influenza Vaccine Evaluation in Kidney Transplant Recipients(AdVEnTR)
Brief Title: Adjuvanted Influenza Vaccine Evaluation in Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: UofA - AdVEnTR
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Influenza
Keywords: kidney transplant recipients
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Influenza is an important public health problem. Organ transplant patients are particularly susceptible to severe disease. Also, they shed higher quantities of virus for longer durations, leading to greater contagious potential, thereby potentially serving as nodes of spread in the community. Therefore, improved strategies to prevent influenza in this population is an important public health concern. Standard vaccination is poorly immunogenic post-transplant and new vaccine strategies are needed. Adjuvanted vaccines contain molecules that create a strong local inflammatory response and they attract immune cells to the site of injection, increasing the immunogenicity of the vaccine antigen. Recently seasonal influenza vaccines containing adjuvants have become available in Canada but have only limited information in transplant patients. This randomized trial is designed to assess the immunogenicity of an adjuvanted vaccination strategy compared to a standard vaccine for seasonal influenza in a cohort of adult organ transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Adult kidney transplant recipients Greater than 3 months post-transplant

Exclusion Criteria:

Has already received influenza vaccination for 2012-2013 season Egg allergy Previous life-threatening reaction to influenza vaccine (i.e. Guillain Barre Syndrome) Ongoing therapy for rejection Febrile illness in the past two weeks Unable to provide informed consent Unable to comply with study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult kidney tranplant recipients
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada